CLINICAL TRIAL: NCT00226967
Title: Stress, Diurnal Cortisol, and Breast Cancer Survival
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB-12273; 76389 (Other: Stanford University Alternate IRB Approval Number); BRSADJ0006 (Other: OnCore)
Record Dates: First submitted 2005-09-13; First posted 2005-09-27 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2019-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Octreotide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Sandostatin — Calculated per patient
  Other Names: Octreotide; Octreo

SUMMARY:
The purpose of this study is to learn about the effects of stress on hormones, the relationship between these hormones and cancer progression.

DETAILED DESCRIPTION:
The purpose of this study is to investigate stress and tonic activation of diurnal cortisol in aging metastatic breast cancer patients; feedback inhibition & activation of cortisol; and stress-induced phasic activation of cortisol.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of recurrent or metastatic breast cancer.
2. Karnofsky of 70% or greater.
3. Proficient enough in English to be able to take questionnaires and participate in the required tasks.
4. Living within the Greater Bay Area.
5. Age 35 or older .

Exclusion Criteria:

1. Positive supraclavicular lymph nodes as the only metastatic lesion at the time of initial diagnosis.
2. Active cancers within the past 10 years other than breast cancer, basal cell or squamous cell carcinomas of the skin, or in situ cancer of the cervix.
3. Any other serious medical condition that will effect short term survival
4. History of major psychiatric illness for which patient was hospitalized or medicated, with the exception of depression or anxiety
5. A diagnosis of diabetes.

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with recurrent or metastatic breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2002-09-08 (Actual); Primary Completion 2004-11 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Spiegel, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States